CLINICAL TRIAL: NCT05878041
Title: Creation of a Multicenter National Registry for Peripartum Cardiomyopathy: a Wide, Multidisciplinary and Translational Perspective to Achieve Personalized Medicine for a Rare Disease in Women
Brief Title: Creation of a Multicenter National Registry for Peripartum Cardiomyopathy.
Acronym: PPCMREGISTRY
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Collaborators: San Raffaele University Hospital, Italy (Other); San Giuseppe Moscati Hospital (Other)
Responsible Party: Principal Investigator, Cinzia Perrino, Associate Professor of Cardiology, Federico II University
Other Study IDs: PNRR-MR1-2022-12376858
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Peripartum Cardiomyopathy
MeSH Terms: conditions — Peripartum Cardiomyopathy | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cells (PBMCs) and serum will be profiled by whole exome sequencing (PBMCs), and proteomics, metabolomics or transcriptomics assays serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peripartum cardiomyopathy: Diagnosis of Peripartum cardiomyopathy (PPCM) will be defined according to the ESC guidelines as: (i) the development of the disease in the last month of pregnancy or within 5 months of delivery; (i) absence of an identifiable cause of heart failure; (iii) absence of recognizable heart disease before the last month of pregnancy; (iv) left ventricle systolic dysfunction demonstrated by classical echocardiographic criteria.
  Interventions: Diagnostic Test: Molecular and genetic screening
- Healthy pregnant volunteers: Healthy pregnant women
  Interventions: Diagnostic Test: Molecular and genetic screening

INTERVENTIONS:
Diagnostic Test: Molecular and genetic screening — Molecular and genetic screening

SUMMARY:
Peripartum cardiomyopathy (PPCM) is a rare, severe and potentially life-threatening disorder of largely unknown etiology and pathophysiology, with unexplained geographical differences and heterogeneous presentation. Investigators hypothesize that a network-based multidisciplinary strategy integrating clinical and molecular phenotyping of PPCM patients might anticipate diagnosis, optimize treatments, and identify novel mechanisms to achieve the unmet goal of personalized medicine.

DETAILED DESCRIPTION:
Specific aims of this study are: a) to create a multicenter pilot registry of PPCM in different areas in Italy to assess incidence and prevalence of this rare disease, associated comorbidities and risk factors. b) to deeply characterize identified PPCM patients through clinical, imaging, genetic, biochemical, and molecular phenotyping. c) to gain novel mechanistic information on PPCM by performing deep clinical and molecular phenotyping in available biobanks samples of patients with PPCM and healthy controls.

ELIGIBILITY:
Inclusion Criteria

* Development of HF signs or symptoms in the last month of pregnancy or within 5 months of delivery;
* Left ventricle systolic dysfunction demonstrated by classical echocardiographic criteria (LVEF< 45 %) in the last month of pregnancy or within 5 months of delivery.

Exclusion Criteria

* Presence of any identifiable cause of HF;
* Presence of recognizable heart disease before the last month of pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnosis of PPCM will be defined according to the ESC guidelines as: (i) the development of the disease in the last month of pregnancy or within 5 months of delivery; (i) absence of an identifiable cause of heart failure; (iii) absence of recognizable heart disease before the last month of pregnancy; (iv) left ventricle systolic dysfunction demonstrated by classical echocardiographic criteria (Eur Heart J 2018;34: 3165; Eur Heart J 2021; 42: 3599). Like other rare diseases, correct diagnosis of PPCM is mostly based on exclusion criteria; however, the differential diagnosis between PPCM, pre-existing chronic heart failure, and other causes of acute heart failure in the peripartum scenario remains challenging.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-02-19 (Estimated); Study Completion 2026-05-19 (Estimated)

PRIMARY OUTCOMES:
Death or hospitalization due to heart failure | 0-6 months
  Death or hospitalization due to heart failure during the follow-up period
Development of significant cardiac arrhythmias | 0-6 months
  New onset sustained supraventricular or ventricular arrhythmias or conduction blocks during the follow-up period

SECONDARY OUTCOMES:
Left ventricular dysfunction | 0-6 months
  Left ventricular % ejection fraction during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Cinzia Perrino, MD pHD, Principal Investigator — Federico II University
Locations (1):
- Federico II University Hospital, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ilardi F, Manzo R, Peretto G, Lanni F, Peano V, Loffredo FS, Masarone D, Gerardi D, di Maio S, Bardi L, Licciardi M, Montali N, Pezzullo E, Di Lorenzo E, Stabile E, Battaglia C, Calanducci M, Bifulco G, Anastasia L, Carusone F, Cascone A, Di Santo M, Cavoretto PI, D'Alconzo D, Palmentieri A, Carotenuto M, Di Spiezio Sardo A, Ioele D, Paolillo R, Polese P, Saccone G, Esposito G, Chieffo A, Perrino C. Clinical presentation and echocardiographic characteristics of women with peripartum cardiomyopathy: Insights from the Italian Multicentre Registry. Int J Cardiol. 2026 Jan 1;442:133866. doi: 10.1016/j.ijcard.2025.133866. Epub 2025 Sep 4. PMID 40914510